CLINICAL TRIAL: NCT03906136
Title: A Randomized, Open Label Multicenter Trial to Investigate the Efficacy of a Treat-to-target (T2T) Treatment Strategy With Secukinumab (AIN457) as a First-line Biologic Compared to a Standard-of-care (SOC) Treatment Over 36 Weeks in Patients With Active Axial Spondyloarthritis (axSpA)
Brief Title: AScalate: Treat-to-target in Axial Spondyloarthritis
Acronym: AScalate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457HDE01; 2018-003882-32 (EudraCT Number)
Record Dates: First submitted 2019-03-26; First posted 2019-04-08 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Axial Spondyloarthritis
Keywords: axial spondyloarthritis; axSpA; treat-to-target; T2T; secukinumab; AIN457; Non-Radiographic Axial Spondyloarthritis; nr-axSpA; Radiographic Axial Spondyloarthritis; r-axSpA
MeSH Terms: conditions — Axial Spondyloarthritis; Non-Radiographic Axial Spondyloarthritis | interventions — secukinumab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREAT-TO-TARGET (T2T) (Experimental): Patients received secukinumab 150 mg subcutaneous (s.c.) weekly until Week 4 (Baseline, Week 1, Week 2, Week 3, Week 4)) and then at Week 8. At Week 12, if ASDAS clinically important improvement was achieved and maintained, patients received treatment up to Week 32 if they maintained the response. If ASDAS clinically important improvement was not achieved, patients received an escalated dose of secukinumab 300 mg s.c. every 4 weeks until Week 20.
  At Week 24, patients who were receiving secukinumab 300 mg, and achieved ASDAS clinically important improvement, continued treatment up to Week 32. If patients did not achieve ASDAS clinically important improvement, they were switched to adalimumab biosimilar (Hyrimoz®) 40 mg s.c. every 2 weeks until Week 34.
  Each patient was treated for a maximum of 36 weeks (last dose of secukinumab at Week 32, last dose of adalimumab biosimilar (Hyrimoz®) at Week 34).
  Interventions: Biological: Secukinumab/Adalimumab-Biosimilar
- Standard-of-care (SOC) (Active Comparator): Patients received SOC treatment according to local practice standards by their treating rheumatologist following latest treatment recommendations with NSAIDs as the first-choice drug treatment and disease-modifying anti-rheumatic drugs (DMARDs) for patients with active disease despite the use (or intolerance/contraindication) of NSAIDs.
  Interventions: Other: Standard-of-care

INTERVENTIONS:
Biological: Secukinumab/Adalimumab-Biosimilar — Secukinumab 150 mg, s.c. Secukinumab 300 mg, s.c. Adalimumab biosimilar 40 mg, s.c.
  Arms: TREAT-TO-TARGET (T2T)
Other: Standard-of-care — Treatment according to local practice standards by the rheumatologist following latest treatment recommendations with NSAIDs as the first-choice drug treatment and DMARDs for patients with active disease despite the use (or intolerance/contraindication) of NSAIDs.
  Arms: Standard-of-care (SOC)

SUMMARY:
This was a randomized, parallel-group, open-label, multicenter study in patients with active axSpA. The aim of the study was to demonstrate that the efficacy of a T2T approach (with secukinumab as a first-line biologic) was superior to a SOC approach in terms of achieving strong clinical efficacy in patients with active axSpA who were naïve to biological therapy and who had an inadequate response to prior non-steroidal anti-inflammatory drug (NSAID) treatment.

DETAILED DESCRIPTION:
The study included an 8-week Screening period, a 36-week treatment period, and a 20-week safety follow-up period. Neither investigators nor patients were blinded. The primary endpoint was the percentage of patients achieving an ASAS40 response at Week 24. At Baseline, patients were randomized equally to one of two treatment groups (T2T or SOC).

Patients were evaluated every 12 weeks from Baseline through to Week 36. Safety evaluations were included in the regular visits; in addition, a safety follow-up visit was performed 20 weeks after the last study visit (i.e. Week 36) and took place at Week 56 for patients completing the study according to the protocol.

Patients assigned to the SOC treatment group received SOC treatment at the discretion of the investigator in accordance with current clinical practice.

Patients assigned to the T2T treatment group received first line biological treatment with secukinumab 150 mg. Responders were defined as those patients with an ASDAS clinically important improvement of ≥ 1.1.

At week 12 responders continued secukinumab 150 mg, whereas treatment was escalated to 300 mg for non-responders.

At week 24, disease activity was assessed again. Patients who qualify as responders continued the treatment they received prior (either secukinumab 150 mg or 300 mg), patients who were non-responders at week 24 were escalated in treatment: patients who received secukinumab 300 mg before were switched to Adalimumab, and patients who received secukinumab 150mg before were escalated to secukinumab 300mg.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Axial Spondyloarthritis, axSpA (either Non-Radiographic Axial Spondyloarthritis or Radiographic Axial Spondyloarthritis) fulfilling the Ankylosing Spondyloarthritis International Society classification criteria for axSpA
* Active disease as defined by having an Ankylosing Spondylitis Disease Activity Score ≥ 2.1 at Screening and Baseline despite concurrent Non-Steroidal Anti-Inflammatory Drug (NSAID) therapy, or intolerance/contraindication to NSAIDs.
* Objective signs of inflammation at Screening as defined by: Magnetic Resonance Imaging (MRI) of sacroiliac joints performed up to 3 months prior to screening showing acute inflammatory lesion(s), OR elevated quick C-reactive Protein (CRP) (> 5 mg/L), OR MRI showing acute inflammatory lesion(s) in the sacroiliac joints and spine performed during screening period.
* Inadequate response to NSAIDs

Exclusion Criteria:

* Previous exposure to secukinumab or other biologic drug directly targeting Interleukin(IL)-17 or IL-17 receptor.
* Patients who have previously been treated with Tumor Necrosis Factor Alpha inhibitors (investigational or approved).
* Patients treated with any cell-depleting therapies.
* Active ongoing inflammatory diseases or underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal conditions, which in the opinion of the investigator immunosuppressed the patient and/or places the patient at unacceptable risk for participation in an immunomodulatory therapy.
* History of clinically significant liver disease or liver injury
* History of renal trauma, glomerulonephritis, or patients with one kidney only, or a serum creatinine level exceeding 1.8 mg/dL (159.12 μmol/L).
* Active systemic infections during the last 2 weeks (exception: common cold) prior to randomization.
* History of ongoing, chronic or recurrent infectious disease or evidence of tuberculosis (TB) infection
* Patients positive for human immunodeficiency virus, hepatitis B or hepatitis C
* Life vaccinations within 6 weeks prior to Baseline or planned vaccination during study participation until 12 weeks after last study treatment administration.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (38):
- France (13):
  - Novartis Investigative Site, Nice, Cedex1
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Caluire-et-Cuire
  - Novartis Investigative Site, Chambray-lès-Tours
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, La Roche-sur-Yon
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Orléans
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (25):
  - Novartis Investigative Site, Bad Doberan
  - Novartis Investigative Site, Bad Pyrmont
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Ehringshausen
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Freiberg
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Ratingen
  - Novartis Investigative Site, Rendsburg
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Ulm

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Poddubnyy D, Hammel L, Heyne M, Veit J, Jentzsch C, Baraliakos X. Treat-to-target strategy with secukinumab as a first-line biological disease modifying anti-rheumatic drug compared to standard-of-care treatment in patients with active axial spondyloarthritis: protocol for a randomised open-label phase III study, AScalate. BMJ Open. 2020 Sep 30;10(9):e039059. doi: 10.1136/bmjopen-2020-039059. PMID 32998926
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1836

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included an 8-week Screening period.
Groups:
- Treat-to-Target (T2T): Treat To Target approach with secukinumab as first line biologic
- Standard-of-care (SOC): Patients received treatment according to local practice standards by their treating physician following the current treatment recommendations
Period: Overall Study
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Started | 155 | 149
Completed | 143 | 138
Not Completed | 12 | 11
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 7 | 4
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 3 | 7

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) comprised all patients to whom study treatment/reference treatment has been assigned by randomization. According to the intent to treat principle, patients were analyzed according to the treatment they have been assigned to during the randomization procedure.
Groups:
- Treat-to-Target (T2T): Participants received secukinumab at a dose of 150 milligrams (mg) as subcutaneous (s.c.) injection at 150 mg dose at Baseline, Week 1, 2, 3, 4 and 8. From Week 12, only responders continued to receive 4-weekly doses until Week 32 if they maintained the response. In the event these patients experienced a loss of response from Week 24, they were escalated to secukinumab 300 mg s.c. every 4 weeks until Week 32.
  Patients who were non-responders at Week 12 received 4-weekly secukinumab 300 mg s.c. until Week 24. From Week 24, only responders continued to receive 4-weekly secukinumab 300 mg s.c. until Week 32. Patients who were non-responders to secukinumab 300 mg at Week 24 received biweekly adalimumab biosimilar 40 mg s.c. until Week 34.
- Total: Total of all reporting groups
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC) | Total
Number analyzed (Participants) | 155 | 149 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 149 | 144 | 293
  >=65 years | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.0 (12.03) | 38.6 (12.17) | 39.3 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 51 | 110
  Male | 96 | 98 | 194
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 0 | 1 | 1
  White | 128 | 114 | 242
  More than one race | 0 | 1 | 1
  Other | 26 | 33 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving an ASAS40 Response at Week 24
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consists of 4 domains measured on visual analog scales (VAS): 1. Patient's global assessment; 2. Patient's assessment of back pain; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). ASAS40 response is defined as an improvement of ≥40% and ≥2 units on a scale of 0 - 10 in at least three of the four ASAS domains and no worsening at all in the remaining domain. A score of 0 indicates less severity; a score of 10 indicates more severity. Percentage was calculated from a logistic regression model: logit(proportion) = treatment + baseline quick C-reactive protein (CRP) + baseline weight.
Time Frame: Baseline, Week 24
Population: Full Analysis Set (FAS): The FAS comprised all patients to whom study treatment/reference treatment was assigned by randomization. Data represent the number of patients with non-missing response at the specified visit.
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 144 | 139
Percentage of participants | 40.1 | 49.2
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.119, Regression, Logistic; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.43 to 1.10]

2. Secondary Outcome: Percentage of Patients Achieving an ASAS40 Response at Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 147 | 143
Percentage of participants | 34.0 | 46.6
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.37 to 0.95]

3. Secondary Outcome: Percentage of Patients Achieving ASAS20 Response
Description: Assessment of SpondyloArthritis International Society criteria (ASAS) consist of 4 domains measured on visual analog scales (VAS): 1. Patient's global assessment; 2. Patient's assessment of back pain; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI). ASAS20 response is defined as an improvement of ≥20% and ≥1 unit on a scale of 0 - 10 in at least three of the four ASAS domains and no worsening at all in the remaining domain. A score of 0 indicates less severity; a score of 10 indicates more severity. Percentage was calculated from a logistic regression model: logit(proportion) = treatment + baseline quick C-reactive protein (CRP) + baseline weight.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 147 | 143
Percentage of participants
  Week 12 n=147,143 | 51.8 | 60.1
  Week 24 n=144,139: number analyzed (Participants) | 144 | 139
  Week 24 n=144,139 | 62.1 | 65.3
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.154, Regression, Logistic; Odds Ratio (OR) = 0.71, 95% CI 2-sided [0.45 to 1.14]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.562, Regression, Logistic; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.54 to 1.39]

4. Secondary Outcome: Percentage of Patients Achieving ASAS Partial Remission
Description: Assessment of SpondyloArthritis International Society criteria (ASAS): 6 domains (4 main; 2 additional assessment domains): 1. Patient's global assessment measured on a visual analog scale (VAS); 2. Patient's assessment of back pain, measured on a VAS; 3. Function represented by Bath Ankylosing Spondylitis Functional Index (BASFI) average of 10 questions as measured by VAS; 4. Inflammation represented by mean duration and severity of morning stiffness, on the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) as measured by VAS; 5. Spinal mobility represented by the Bath Ankylosing Spondylitis Metrology Index (BASMI) lateral spinal flexion assessment; 6. C-reactive protein (CRP, acute phase reactant).
  ASAS partial remission: a value not above 2 units in each of the four main domains on a scale of 10. Higher score on VAS = higher severity. Percentage calculated from a logistic regression model: logit(proportion) = treatment + baseline quick CRP + baseline weight.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 149 | 143
Percentage of participants
  Week 12 n=149, 143 | 18.2 | 29.0
  Week 24 n=146,139: number analyzed (Participants) | 146 | 139
  Week 24 n=146,139 | 22.8 | 28.5
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.32 to 0.94]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.264, Regression, Logistic; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.44 to 1.25]

5. Secondary Outcome: Percentage of Patients Meeting the Ankylosing Spondylitis Disease Activity Score (ASDAS) Definition of Inactive Disease
Description: Parameters used for the ASDAS include spinal pain (Bath Ankylosing Spondylitis Disease Activity Index, BASDAI question 2), the patient's global assessment of disease activity, peripheral pain/swelling (BASDAI question 3), duration of morning stiffness (BASDAI question 6) and C-reactive Protein or Erythrocyte Sedimentation Rate).
  The 3 values selected to separate disease activity states were < 1.3 between inactive disease and low disease activity, < 2.1 between low disease activity and high disease activity, and > 3.5 between high disease activity and very high disease activity. Selected cutoffs for improvement scores were a change of ≥ 1.1 unit for "minimal clinically important improvement" and a change of ≥ 2.0 units for "major improvement". Percentage was calculated from a logistic regression model: logit(proportion) = treatment + baseline ASDAS + baseline weight.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 151 | 141
Percentage of participants
  Week 12 n=151,141 | 19.8 | 33.3
  Week 24 n=146,136: number analyzed (Participants) | 146 | 136
  Week 24 n=146,136 | 18.8 | 33.0
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.008, Regression, Logistic; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.29 to 0.83]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.005, Regression, Logistic; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.28 to 0.80]

6. Secondary Outcome: Percentage of Patients With ASDAS Major Improvement
Description: as for outcome 5
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 151 | 141
Percentage of participants
  Week 12 n=151,141 | 19.8 | 25.6
  Week 24 n=146,136: number analyzed (Participants) | 146 | 136
  Week 24 n=146,136 | 18.6 | 27.1
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.263, Regression, Logistic; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.40 to 1.28]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.103, Regression, Logistic; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.34 to 1.10]

7. Secondary Outcome: Percentage of Patients With ASDAS Low Disease Activity
Description: as for outcome 5
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 151 | 141
Percentage of participants
  Week 12 n=151,141 | 46.5 | 57.7
  Week 24 n=146,136: number analyzed (Participants) | 146 | 136
  Week 24 n=146,136 | 52.4 | 57.2
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.055, Regression, Logistic; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.40 to 1.01]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.409, Regression, Logistic; Odds Ratio (OR) = 0.82, 95% CI 2-sided [0.52 to 1.31]

8. Secondary Outcome: Percentage of Patients Achieving the Bath Ankylosing Spondylitis Disease Activity Index Response 50% (BASDAI 50) at Week 12 and Week 24
Description: The BASDAI consists of a 0 through 10 scale (0 being no problem and 10 being the worst problem, captured as a continuous VAS), which is used to answer 6 questions pertaining to the 5 major symptoms of the disease. BASDAI 50 response is defined as at least 50% improvement (decrease) in total BASDAI score.
Time Frame: Baseline, Weeks 12 and 24
Population: Full Analysis Set (FAS): The FAS comprised all patients to whom study treatment/reference treatment was assigned by randomization.
Measure: Number; unit: Percentage of participants
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
Percentage of participants
  Week 12 | 38.0 | 42.0
  Week 24 | 42.5 | 42.2
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.477, Regression, Logistic; Odds Ratio (OR) = 0.85, 95% CI 2-sided [0.53 to 1.34]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.968, Regression, Logistic; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.63 to 1.61]

9. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI)
Description: The Bath Ankylosing Spondylitis Functional Index (BASFI) is a set of 10 questions designed to determine the degree of functional limitation in those patients with AS. The 10 questions were chosen with major input from patients with AS. The first 8 questions consider activities related to functional anatomy. The final 2 questions assess the patients' ability to cope with everyday life. A 0 through 10 scale (captured as a continuous VAS) is used to answer the questions. The mean of the 10 scales gives the BASFI score - a value between 0 and 10. A higher score on the VAS signifies higher severity.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
Scores on a scale
  Week 12: number analyzed (Participants) | 153 | 144
  Week 12 | -1.69 [-2.01 to -1.37] | -1.99 [-2.31 to 1.66]
  Week 24: number analyzed (Participants) | 148 | 140
  Week 24 | -1.97 [-2.28 to 1.65] | -2.33 [-2.66 to 2.01]
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.205, Regression, Logistic; Odds Ratio (OR) = 0.30, 95% CI 2-sided [-0.16 to 0.75]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.108, Regression, Logistic; Odds Ratio (OR) = 0.37, 95% CI 2-sided [-0.08 to 0.82]

10. Secondary Outcome: Change From Baseline in Bath Ankylosing Spondylitis Metrology Index (BASMI)
Description: BASMI measures the range of motion based on five clinical measurements: 1) cervical rotation, 2) tragus to wall distance, 3) lumbar side flexion, 4) lumbar flexion (modified Schober's) and 5) intermalleolar distance. BASMI 0 = indicates mild disease involvement, 1 = moderate disease, and 2 = severe disease involvement. The results for cervical rotation and lumbar side flexion are the means of the left and right measurements. Scoring range 0-10. The higher the BASMI score, the more severe was the subject's limitation of movement.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
Scores on a scale
  Week 12: number analyzed (Participants) | 150 | 144
  Week 12 | -0.32 [-0.44 to -0.20] | -0.38 [-0.50 to -0.27]
  Week 24: number analyzed (Participants) | 148 | 135
  Week 24 | -0.41 [-0.55 to -0.27] | -0.35 [-0.50 to -0.21]
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.525, Mixed Models Analysis; Mean Difference (Net) = 0.06, 95% CI 2-sided [-0.12 to 0.23]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.577, Mixed Models Analysis; Mean Difference (Net) = -0.06, 95% CI 2-sided [-0.25 to 0.14]

11. Secondary Outcome: Change From Baseline in Chest Expansion
Description: Chest expansion is measured as the cervical rotation angle (in degrees).
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: degrees
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
degrees
  Week 12: number analyzed (Participants) | 150 | 144
  Week 12 | 0.46 [-0.54 to 1.46] | 1.35 [0.33 to 2.38]
  Week 24: number analyzed (Participants) | 147 | 135
  Week 24 | 0.47 [0.05 to 0.88] | 0.57 [0.14 to 1.00]
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.220, Mixed Models Analysis; Odds Ratio (OR) = -0.89, 95% CI 2-sided [-2.32 to 0.54]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.745, Regression, Logistic; Median Difference (Net) = -0.10, 95% CI 2-sided [-0.70 to 0.50]

12. Secondary Outcome: Change From Baseline in the ASQoL (Ankylosing Spondylitis Quality of Life Instrument)
Description: The Ankylosing Spondylitis Quality of Life scores (ASQoL) is a self-administered questionnaire designed to assess health-related quality of life in adult patients with Ankylosing Spondylitis. The ASQoL contains 18 items with a dichotomous yes/no response option. A single point is assigned for each "yes" response and no points for each "no" response resulting in overall scores that range from 0 (least severity) to 18 (highest severity). As such, lower score indicate better quality of life. Items include an assessment of mobility/energy, self-care and mood/emotion. The recall period is "at the moment," and the measure requires approximately 6 minutes to complete.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
Scores on a scale
  Week 12: number analyzed (Participants) | 150 | 141
  Week 12 | -3.52 [-4.13 to 2.91] | -3.39 [-4.02 to 2.76]
  Week 24 | -4.21 [-4.88 to 3.53] | -3.84 [-4.53 to 3.15]
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.768, Mixed Models Analysis; Mean Difference (Net) = -0.13, 95% CI 2-sided [-1.01 to 0.74]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.451, Mixed Models Analysis; Mean Difference (Net) = -0.37, 95% CI 2-sided [-1.34 to 0.60]

13. Secondary Outcome: Change From Baseline in ASAS-HI (Ankylosing Spondyloarthritis International Society Health Index)
Description: The ASAS-HI is a disease-specific questionnaire that was developed based on the comprehensive International Classification of Functioning, Disability and Health Core Set (also known as the ICF Core Set) for AS. The ASAS HI is a linear composite measure and contains 17 items (dichotomous response option: "I agree" and "I do not agree"), which cover most of the ICF Core Set. The ASAS HI contains items addressing categories of pain, emotional functions, sleep, sexual function, mobility, self-care, and community life. The total sum of the ASAS HI ranges from 0 to 17, with a lower score indicating a better health status. In addition, the Environmental Factor (EF) Item Set contains items addressing categories of support/relationships, attitudes and health services. The EF Item Set contains 9 dichotomous items with an identical response option but without a sum score because of its multidimensional nature.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
Scores on a scale
  Week 12: number analyzed (Participants) | 150 | 143
  Week 12 | -2.55 [-3.05 to 2.05] | -2.81 [-3.32 to 2.30]
  Week 24: number analyzed (Participants) | 147 | 139
  Week 24 | -3.24 [-3.77 to 2.72] | -3.07 [-3.61 to 2.54]
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.477, Mixed Models Analysis; Mean Difference (Net) = 0.26, 95% CI 2-sided [-0.46 to 0.97]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.660, Mixed Models Analysis; Mean Difference (Net) = -0.17, 95% CI 2-sided [-0.92 to 0.58]

14. Secondary Outcome: Change From Baseline in Global Disease Assessment (Patient)
Description: The patient's global assessment of disease activity was performed using a 100 mm (visual analog scale) VAS, ranging from not severe (0 mm) to very severe (100 mm), in response to the question, "How active was your disease on average during the last week?" A higher score indicates more disease activity.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
Scores on a scale
  Week 12: number analyzed (Participants) | 153 | 143
  Week 12 | -2.95 [-3.38 to 2.52] | -3.12 [-3.56 to 2.68]
  Week 24: number analyzed (Participants) | 148 | 139
  Week 24 | -3.27 [-3.69 to 2.85] | -3.48 [-3.92 to 3.05]
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 12; Test type: Superiority; p = 0.586, Mixed Models Analysis; Mean Difference (Net) = 0.17, 95% CI 2-sided [-0.45 to 0.79]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.491, Mixed Models Analysis; Median Difference (Net) = 0.21, 95% CI 2-sided [-0.39 to 0.82]

15. Secondary Outcome: Change From Baseline in Global Disease Assessment (Physician)
Description: The physician's global assessment of disease activity was performed using a 100 mm VAS, ranging from not severe (0 mm) to very severe (100 mm), in response to the question, "Considering all the ways the disease affects your patient, draw a line on the scale for how well his or her condition is today." To enhance objectivity, the physician must not be aware of the specific patient's global assessment of disease activity when performing his own assessment on that patient. A higher score indicates more disease activity.
Time Frame: Baseline, Weeks 12 and 24
Population: as for outcome 8
Measure: Least Squares Mean (90% Confidence Interval); unit: Scores on a scale
Arm/Group | Treat-to-Target (T2T) | Standard-of-care (SOC)
Number analyzed (Participants) | 155 | 149
Scores on a scale
  Week 12: number analyzed (Participants) | 153 | 143
  Week 12 | -32.46 [-35.98 to 28.94] | -36.96 [-40.60 to 33.31]
  Week 24: number analyzed (Participants) | 148 | 149
  Week 24 | -35.81 [-39.34 to 32.28] | -38.54 [-42.19 to 34.89]
Statistical Analysis 1: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Test type: Superiority — Week 12; p = 0.082, Mixed Models Analysis; Mean Difference (Net) = 4.49, 95% CI 2-sided [-0.58 to 9.56]
Statistical Analysis 2: Comparison: Treat-to-Target (T2T) vs Standard-of-care (SOC); Week 24; Test type: Superiority; p = 0.292, Mixed Models Analysis; Median Difference (Net) = 2.73, 95% CI 2-sided [-2.35 to 7.81]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were reported from first dose of study treatment until end of study treatment plus 20 weeks up to approximately 56 weeks.
Description: The safety set included all patients who received at least one dose of study treatment. AEs are reported according to the actual treatment received when AE started. As Secukinumab 150 mg could also had been provided in the Standard-of-Care arm, the number of patients at risk exceeds the number of patients enrolled in the T2T arm. For AEs that occurred while on other treatment in the SoC arm, the specific treatment information was not collected, and AEs summarized under one arm.
Groups:
- Secukinumab 150 mg: Secukinumab 150 mg
- Secukinumab 300 mg: Secukinumab 300 mg
- Adalimumab 40 mg: Adalimumab 40 mg
- Other Treatment: Other treatment included concomitant and rescue medications other than study drugs.
- Overall: Overall
Arm/Group | Secukinumab 150 mg | Secukinumab 300 mg | Adalimumab 40 mg | Other Treatment | Overall
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/92 | 0/116 | 0/128 | 0/303
Serious Adverse Events (participants affected / at risk) | 10/190 | 4/92 | 5/116 | 8/128 | 16/303
Other Adverse Events (participants affected / at risk) | 69/190 | 38/92 | 35/116 | 36/128 | 98/303
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg (N=190) | Secukinumab 300 mg (N=92) | Adalimumab 40 mg (N=116) | Other Treatment (N=128) | Overall (N=303)
Angina pectoris (Cardiac disorders) | 1 | 1 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Immunisation reaction (Immune system disorders) | 1 | 0 | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 1 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 150 mg (N=190) | Secukinumab 300 mg (N=92) | Adalimumab 40 mg (N=116) | Other Treatment (N=128) | Overall (N=303)
Diarrhoea (Gastrointestinal disorders) | 16 | 9 | 8 | 11 | 24
Nausea (Gastrointestinal disorders) | 12 | 6 | 3 | 7 | 14
Fatigue (General disorders) | 7 | 3 | 6 | 5 | 12
Nasopharyngitis (Infections and infestations) | 24 | 13 | 7 | 10 | 31
Respiratory tract infection (Infections and infestations) | 10 | 3 | 3 | 3 | 10
Upper respiratory tract infection (Infections and infestations) | 10 | 6 | 6 | 3 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 3 | 0 | 8
Headache (Nervous system disorders) | 12 | 7 | 7 | 6 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/36/NCT03906136/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT03906136/SAP_001.pdf